CLINICAL TRIAL: NCT03032770
Title: Early Prediction of Placenta Accreta by 2 Dimensional Transvaginal Ultrasound and Color Doppler
Brief Title: Early Prediction of Placenta Accreta by Ultrasound and Color Doppler
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, clinical professor, Assiut University
Other Study IDs: USPA
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- placenta accreta: Having at least one sign suggestive of placenta accreta
  Interventions: Device: two-dimensional ultrasound and color Doppler
- normal placenta: Never having any of the signs suggestive of placenta accreta
  Interventions: Device: two-dimensional ultrasound and color Doppler

INTERVENTIONS:
Device: two-dimensional ultrasound and color Doppler — the eligible participants will be searched for signs suggestive of placenta accreta; low implantation of the gestational sac (<4cm from the external os), presence of placental lakes, Disruption of placental-myometrial interface and trophoblast overlapping a uterine scar by 2 dimensional transvaginal ultrasound and Intraplacental dilated vessels, turbulent blood flows and greatly increased periplacental vascularity by Doppler ultrasound by level II sonographer and co-investigator under his supervision using ultrasound device.

SUMMARY:
Placenta accreta is a substantially life threatening condition and one of the causes of maternal morbidity and mortality in the world. According to study done in United Kingdom, The estimated incidence of placenta accreta/increta/percreta was 1.7 per 10,000 maternities overall and 577 per 10,000 in women with both a previous cesarean delivery and placenta previa. in a tertiary south Italian center, The incidence increased from 0.12% during the 1970s, to 0.31% during the 2000s.While in United States of America, the prevalence of placenta accreta was 3.7 per 1000 deliveries.

ELIGIBILITY:
Inclusion Criteria:

1. Low implantation of the gestational sac (<4 cm from external os) by transvaginal ultrasound
2. Presence of placental lakes by transvaginal ultrasound
3. Disruption of placental-myometrial interface by transvaginal ultrasound
4. Trophoblast overlapping a uterine scar (Cesarean section, myomectomy) by transvaginal ultrasound
5. Intraplacental dilated vessels by Doppler ultrasound
6. Turbulent blood flows by Doppler ultrasound
7. Greatly increased periplacental vascularity by Doppler ultrasound

Exclusion Criteria:

a) Cases far away from our hospital and expected to be lost to be followed. b) Pregnant women who will refuse to Participate

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: first trimester pregnancy between 11 weeks and 13 weeks.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Confirmation of occurrence of placenta accreta during delivery. | duration of pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided